CLINICAL TRIAL: NCT03187366
Title: EID: Using Community Ecology Theory to Predict the Effects of Agricultural Expansion and Intensification on Infections of Humans: Implications for Sustainable Agriculture
Brief Title: Schistosomiasis in Senegal
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Notre Dame (Other)
Collaborators: Biomedical Research Center EPLS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01TW010286 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Schistosomiasis
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Status quo (No Intervention): Status quo pesticide use
- Low risk (Active Comparator): Villages shifted to low risk pesticides that don't kill prawns
  Interventions: Other: Bottom-up intervention
- No agrochemicals (Experimental): Villages that eliminate agrochemicals
  Interventions: Other: Bottom-up intervention

INTERVENTIONS:
Other: Bottom-up intervention — Some interventions are bottom-up, where we manipulate the resources of snails and some are top-down, where we manipulate the predators of snails.
  Other Names: Top-down intervention
  Arms: Low risk; No agrochemicals

SUMMARY:
Schistosomiasis is a flatworm transmitted from freshwater snails to humans in the tropics. In addition to this infectious disease, tropical developing countries are faced with malnutrition. We propose to alter pesticide and compost use to reduce schistosomiasis and maintain or even improve crop production.

DETAILED DESCRIPTION:
We propose two types of manipulations. Bottom-up manipulations will affect snail resources, whereas top-down manipulations will affect snail predators. For the bottom-up manipulations, we will clear schistosoma infections in school children, then remove the primary habitat for snails, the submerged macrophyte Ceratophyllum demersum (with proper unmanipulated controls), compost it, apply it to crops, and then quantify reinfection rates and crop yields. The second bottom-up manipulation will be to clear schistosoma infections in school children, apply three agrochemical treatments (status quo control, shift to lower risk herbicides, or eliminate herbicides and fertilizers), and then quantify reinfection rates and crop yields. Farmers will be compensated for any loss in yields. For the top-down manipulations, every village will receive prawns that depredate snails. We will clear schistosoma infections in school children, apply three agrochemical treatments (status quo control, shift to lower risk insecticides that don't kill prawns, or eliminate insecticides), and then quantify reinfection rates and crop yields. Farmers will be compensated for any loss in yields.

ELIGIBILITY:
Inclusion Criteria:

* School age children

Exclusion Criteria:

* Non-school age children

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1477 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Schistosomiasis reinfection rate | One year
  Schistosomiasis reinfection rate

SECONDARY OUTCOMES:
Crop yields | One year
  Crop yields

CONTACTS AND LOCATIONS:
Overall Officials: Jason R Rohr, PhD, Principal Investigator — University of South Florida, Department of Integrative Biology
Locations (1):
- Espoir Pour La Santé (EPLS), Saint-Louis, Senegal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rohr JR, Sack A, Bakhoum S, Barrett CB, Lopez-Carr D, Chamberlin AJ, Civitello DJ, Diatta C, Doruska MJ, De Leo GA, Haggerty CJE, Jones IJ, Jouanard N, Lund AJ, Ly AT, Ndione RA, Remais JV, Riveau G, Schacht AM, Seck M, Senghor S, Sokolow SH, Wolfe C. A planetary health innovation for disease, food and water challenges in Africa. Nature. 2023 Jul;619(7971):782-787. doi: 10.1038/s41586-023-06313-z. Epub 2023 Jul 12. PMID 37438520